CLINICAL TRIAL: NCT06151743
Title: Neoadjuvant Therapy With Toripalimab Combined With Cetuximab and Platinum for Resectable Locally Advanced Hypopharyngeal Cancer
Brief Title: Neoadjuvant PD-1 Inhibitor Combined With Cetuximab and Platinum in Resectable Locally Advanced Hypopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPC-SCCHN
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-11

CONDITIONS: Locally Advanced Hypopharyngeal Carcinoma
MeSH Terms: interventions — toripalimab; Cetuximab; Platinum; Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy+Surgery+Adjuvant therapy (Experimental): Participants receive three cycles of neoadjuvant therapy (toripalimab+cetuximab+platinum), followed by radical surgery. After surgery, participants receive radiotherapy or chemoradiotherapy according to the pathological results of the operation.
  Interventions: Drug: three cycles (toripalimab + cetuximab + platinum); Procedure: Radical surgery; Radiation: Radiotherapy or chemoradiotherapy

INTERVENTIONS:
Drug: three cycles (toripalimab + cetuximab + platinum) — Cetuximab 250 mg/m2 i.v. qw (first loading dose 400 mg/m2) for nine doses; Toripalimab 240 mg/m2 i.v. d1, q21d, three cycles; Cisplatin 25 mg/m2 i.v. d1-3, q21d, three cycles or Carboplatin AUC 5 i.v. d1, q21d, three cycles (patients with cisplatin contraindications or renal impairment after cisplatin use).
  Other Names: Toripalimab + Cetuximab + Platinum
Procedure: Radical surgery — The attending physician should select the appropriate surgical treatment and try to perform radical laryngeal preservation surgery for patients with tumor retraction after induction therapy. Patients who cannot preserve laryngeal function due to tumor load need to undergo total laryngeal resection. According to the scope of pharyngectomy, the surgical treatments include partial laryngopharyngectomy, total laryngectomy and partial pharyngectomy, total laryngopharyngectomy, and total pharyngo-laryngo-esophagectomy. Cervical lymph node dissection was performed when necessary.
Radiation: Radiotherapy or chemoradiotherapy — 1. Using intensity-modulated radiotherapy (IMRT) technology, the dose of radiotherapy is determined according to whether there are adverse prognostic factors in the postoperative pathology, including positive margins, extracapsular invasion of lymph nodes, primary pT3 or T4, N2 lymph node lesions, peripheral nerve invasion, vascular/lymphatic infiltration.
     Primary site: residual GTV or tumor bed dose 60-70Gy: 1.8-2.12 Gy / fraction. Cervical lymph nodes or lymphatic drainage area: 56-70 Gy: 1.7-2.12 Gy / fraction.
  2. Postoperative adjuvant concurrent chemotherapy regimen:
  Cisplatin 25mg/m2 i.v. d1-3, d22-24 or Carboplatin AUC 5 i.v. d1, d22 (if cisplatin contraindications).

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of immunotherapy combined with cetuximab and platinum neoadjuvant therapy in patients with resectable locally advanced hypopharyngeal cancer. Participants will receive three cycles of TPC neoadjuvant therapy (toripalimab+ cetuximab + platinum), radical surgery (laryngeal preservation surgery if possible), and sequential (chemo)radiotherapy treatment after surgery. This trial aims to answer the following questions:

1. pCR rate
2. MPR rate, ORR, LPR/DFS/OS rare at 1 and 2 years
3. Safety and quality of life

DETAILED DESCRIPTION:
The standard treatment for patients with resectable hypopharyngeal carcinoma is surgery plus postoperative adjuvant radiotherapy or chemoradiotherapy. Growing evidence shows that neoadjuvant therapy may significantly increase pCR in locally advanced SCCHN patients, potentially improving patient survival. The development of drugs, immunotherapy, and targeted therapy has been proven to improve the overall survival of patients with SCCHN significantly, and PD-1 inhibitor combined with cetuximab has also shown promising efficacy in R/M SCCHN. This study explores the effectiveness and safety of immunotherapy combined with cetuximab and platinum neoadjuvant therapy in patients with resectable locally advanced hypopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as hypopharyngeal squamous cell carcinoma;
* Age between 18-75 years;
* Patients with resectable locally advanced hypopharyngeal cancer with T3-4aN0-3bM0 (AJCC 8th) require total laryngectomy;
* Have at least one evaluable target lesion according to RECIST 1.1 criteria.
* No previous treatment for hypopharyngeal carcinoma;
* Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-1;
* Estimated survival ≥ 6 months;
* Normal organ function;
* HBV DNA < 500 IU/mL (or 2500 copies/mL) and HCV RNA negative;
* Signed informed consent;
* Patients who are compliant, willing, and able to follow visiting schedules, treatment plans, laboratory tests, and other research procedures.
* Male and no pregnant female; able to use the contraceptive method during treatment.

Exclusion Criteria:

* Have a history of other cancers in the past five years, except for the following cancers that are cured in the past five years: basal cell carcinoma and squamous cell carcinoma of the skin, early prostate cancer, papillary thyroid cancer, breast ductal carcinoma in situ and cervix carcinoma in situ;
* The target lesion has been treated with radiation therapy or surgery, except for biopsy to confirm the diagnosis of hypopharyngeal carcinoma;
* Previous chemotherapy, immunotherapy, or bio-targeted therapy for the primary tumor;
* Patients who have participated in other clinical trials within four weeks before the trial;
* Any of the following diseases within six months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
* Those with hypertension who cannot be reduced to normal range by antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
* Patients with grade I or above coronary heart disease, arrhythmia (including QTc interval prolongation > 450 ms for men and > 470 ms for women), and cardiac insufficiency.
* Patients with positive urine protein (urine protein test 2 + or above, or 24-hour urine protein quantification >1.0g).
* Patients with severe allergic history or allergic constitution; an active autoimmune disease that may worsen when receiving immunostimulants. Patients with type I diabetes, vitiligo, psoriasis, or diseases of hypothyroidism or hyperthyroidism that do not require immunosuppressive therapy are eligible to participate in the study.
* Subjects requiring systemic therapy with corticosteroids (> 10 mg prednisone or equivalent) or other immunosuppressants within two weeks before the first use of the study drug.
* Previously diagnosed immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) - related disease. hepatitis B virus (HBV) surface antigen positive and HBV-DNA ≥ 500 IU/mL (or 2500 copies/mL), or HCV RNA positive. History of active or previous tuberculosis (TB).
* Patients with a history of psychotropic substance abuse who cannot quit or have mental disorders.
* Vaccination within four weeks before enrollment, except for inactivated vaccine.
* Pregnant or lactating women, those who are in the reproductive period and do not use effective contraception;
* Those whom the investigator deems unsuitable to participate in this trial, such as severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or psychiatric illness (including recent or active suicidal ideation or behavior) or abnormal laboratory tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate after neoadjuvant chemotherapy | Within 3 weeks after surgery
  The pCR rate is defined as the percentage of participants who have no residual tumor cells in the resected primary tumor within 14 weeks after the start of neoadjuvant therapy.

SECONDARY OUTCOMES:
Major pathologic response (MPR) rate | Within 3 weeks after surgery
  MPR rate, defined as no more than 10% of residual viable tumor, evaluated by experienced pathologists.
Objective response rate (ORR) after neoadjuvant therapy | Up to 14 weeks after the start of neoadjuvant therapy
  The ORR is the proportion of patients whose tumor volume was reduced to 30% and sustained for more than 4 weeks as assessed by RECIST 1.1.
1-year and 2-year larynx preservation rate (LPR) | Two years post-radiotherapy
  LPR is the proportion of patients who avoid total laryngectomy. 1-year and 2-year LPR is defined as the probability of larynx preservation for a patient at a given time (1 year and 2 years).
1-year and 2-year disease-free survival (DFS) rate | Two years post-radiotherapy
  DFS is the time from enrollment until radiographic disease progression, local or distant recurrence, or death due to any cause. The 1-year and 2-year DFS rate is the probability of disease-free survival for a patient at a given time (1 year and 2 years).
1-year and 2-year overall survival (OS) rate | Two years post-radiotherapy
  OS is the time from enrollment to death due to any cause. The 1-year and 2-year OS rates are the probability of overall survival for a patient at a given time (1 year and 2 years).
Adverse Effect | One year post-radiotherapy
  Adverse Effect, evaluated by CTCAE V5.0

OTHER OUTCOMES:
Quality of Life Score (QoL) | Two years post-radiotherapy
  Refer to EORTC QLQ-C30 (version 3, version Chinese). After the end of treatment, it is assessed every 3 months (for patients after PD, subsequent quality of life assessment is no longer performed).
Biomarker detection | Two years post-radiotherapy
  Peripheral blood samples and surgical tissue samples are retained for correlation analysis of PD-1/PD-L1 expression levels with efficacy and prognosis and screening for genes or markers related to efficacy and prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Tao, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No